CLINICAL TRIAL: NCT06056856
Title: Anatomical and Functional Outcome of Penile Skin Graft Versus Buccal Mucosal Graft for Urethral Substitution in Long Segment Anterior Urethral Strictures
Brief Title: Anatomical and Functional Outcome of PSG Vs BMG for Urethral Substitution in Long Segment Anterior Urethral Strictures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Anwar, Assistant lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 773
Record Dates: First submitted 2023-08-11; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Anterior Urethral Stricture, Male
Keywords: urethral stricture; urethroplasty; BMG; PSG; penile skin
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Intervention Model Description: Two-arm parallel assignment. The first arm will be operated using penile skin grafts, The second arm will be operated using buccal mucosal grafts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSG group (Active Comparator): The group of patients who will undergo penile skin graft substitituion of long anterior urethral stricture
  Interventions: Procedure: Penile skin graft substituttion urethroplasty
- BMG group (Active Comparator): The group of patients who will undergo buccal mucosal graft substitituion of long anterior urethral stricture
  Interventions: Procedure: Buccal Mucosal Graft substitution urethroplasty

INTERVENTIONS:
Procedure: Penile skin graft substituttion urethroplasty — substitution of long anterior urethral strictures using one-sided dorsal perineal approach
  Arms: PSG group
Procedure: Buccal Mucosal Graft substitution urethroplasty — substitution of long anterior urethral strictures using one-sided dorsal perineal approach
  Arms: BMG group

SUMMARY:
This study aims to compare the penile skin graft and buccal mucosal graft for substitution of long anterior urethral strictures using one-sided dorsal perineal approach.

DETAILED DESCRIPTION:
Since previous studies were:

* Retrospective and very few were prospective randomized studies
* Some studies were done on lichen sclerosis cases that have an adverse effect on the PSG outcome.
* The follow-up duration was longer for PSG patients.
* Stricture length was usually longer for PSG cases.

This study aims to compare the PSG and BMG for substitution of long anterior urethral strictures using one-sided dorsal perineal approach.

The investigators hypothesize that:

❶ Conducting a well-designed prospective, randomized study can help identify which technique is better than the other.

❷ Using the one-side dorsal approach can improve the outcomes of both techniques and identify their advantages and disadvantages.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients with long segment anterior urethral stricture (>2 cm).

Exclusion Criteria:

* Urethro-cutaneous fistula, urethral abscess or diverticulum.
* A scarred and unsalvageable urethral plate or scarred perineum.
* Lichen sclerosis (Balanitis xerotica obliterans).
* Unhealthy/unavailable buccal mucosa.

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
The degree of urethral lumen patency. | through study completion, an average of 1 year.
  Patent urethra as evidenced by uroflowmetry and retrograde urethrography +/- urethroscopy

SECONDARY OUTCOMES:
Lower urinary tract symptoms improvement | 6 months
  lower urinary tract symptoms as assessed by the international prostate symptom score, ranging from 0 to 35, where scores from 0-7 are mild, from 8-19 are moderate, from 20-35 are severe symptoms.
Erectile function assessment | 6 months
  sexual function as assessed by the international index of erectile function-5 questionnaire, ranging from 5-25, where 22-25 is normal, 17-21 is mild ED, 12-16 is mild to moderate ED, 8-11 is moderate ED, and 5-7 is severe ED.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Fahim, professor, Study Director — Urology department, Al-Azhar university, Cairo, Egypt; Mostafa Ezzeldein, professor, Study Chair — Urology department, Al-Azhar university, Cairo, Egypt
Locations (1):
- Al-Azhar urology department, Al-Azhar university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Patients' data sheet, patient consent forms through my E-mail: m0anwar2005@gmail.com
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available after 1 year, and for 2 years.
Access Criteria: My e-mail: m0anwar2005@gmail.com

DOCUMENTS (1):
  • Study Protocol (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/56/NCT06056856/Prot_000.pdf